CLINICAL TRIAL: NCT05043974
Title: Integrative Study of Physiological Changes Induced by a 5-Day Dry Immersion, Used as a Ground-based Model to Mimic Weightlessness: a Pilot Study on 20 Healthy Female Volunteers (DI5-Women Study)
Brief Title: Integrative Study of Physiological Changes Induced by a 5-Day Dry Immersion on 20 Healthy Female Volunteers (DI5-Women)
Acronym: VivalDI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre National d'Etudes Spatiales (Other Government)
Collaborators: European Space Agency (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 20-232; 2021-A00705-36 (Other: ANSM)
Record Dates: First submitted 2021-07-30; First posted 2021-09-14 (Actual); Last update posted 2022-07-21 (Actual); Status verified 2021-09

CONDITIONS: Weightlessness; Weightlessness; Adverse Effect
Keywords: Simulated Microgravity; Weightlessness; Dry immersion; Supportlessness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dry immersion (Experimental): 5 days of dry-immersion.
  Interventions: Other: Dry immersion

INTERVENTIONS:
Other: Dry immersion — Subjects are immersed up to the neck for 5 days in a specially designed bath filled with tap water.

SUMMARY:
Dry immersion (DI) is a ground-based model of prolonged conditions of simulated microgravity. Dry immersion involves immersing the subject in water covered with an elastic waterproof fabric. As a result, the immersed subject, who is freely suspended in the water mass, remains dry. Within a relatively short duration, the model can faithfully reproduce most physiological effects of actual microgravity, including centralization of body fluids, support unloading, and hypokinesia.

The objective of the study is to evaluate the physiological changes induced by 5 days of dry immersion in the female organism. The main physiological systems will be explored before, during and after the 5 days of immersion through a battery of specific tests and measurements. The results will be analyzed by scientists specializing in each field in order to better understand the dry immersion model, to compare its effects with those of the bedrest model and those of spaceflight. The clinical (adverse effects, comfort of subjects) and operational aspects are also part of the secondary objectives of the study.

DETAILED DESCRIPTION:
The space agencies are actively engaged in studying the physiological adaptation to space environment through studies on board the International Space Station (ISS) but also on the ground. Ground-based experiments simulating the effects of weightlessness are used to better understand the mechanisms of physiological adaptation, design and validate the countermeasures. Dry immersion (DI) is a ground-based model of prolonged conditions of simulated microgravity, which has been mainly used in Russia. The past years however, the model has been implemented as well in Europe and expertise in conducting DI studies has been gained in particular in France where a few DI studies have been conducted in the MEDES Space Clinic in Toulouse for CNES (French Space Agency). Dry immersion involves immersing the subject in water covered with an elastic waterproof fabric. As a result, the immersed subject, who is freely suspended in the water mass, remains dry. Within a relatively short duration, the model can faithfully reproduce most physiological effects of actual microgravity, including centralization of body fluids, support unloading, and hypokinesia. Furthermore, physiological changes have been reported in the neuromuscular, skeletal and sensorimotor systems, in fluid electrolyte regulation, in the cardiovascular system, metabolism, blood and immunity, respiration, and thermoregulation. Dry immersion provides a unique opportunity to study the physiological effects of the lack of a supporting structure for the body (a phenomenon called 'supportlessness'). As such, dry immersion is proposed to mimic actual spaceflight in terms of the monotonous environment, posture-motion limitations, hemodynamic changes and hypokinetic effects, support unloading, and decreased proprioceptive input. Immersion studies have so far only been conducted in men and a minority of studies using the bedrest model have included women. Likewise, few studies conducted to date have investigated gender differences in the astronaut population. The small number of female astronauts may be part of the reason why scientific data are lacking to draw valid conclusions about possible gender differences. However, if women currently constitute only about 10% of astronauts, women are and will be more and more represented in crews. Women now constitute 30% of American crews and NASA (US space agency) has announced gender parity for crews on future lunar missions. It is therefore essential to study the physiological changes induced by weightlessness in women, to compare them with those observed in men and to develop efficient countermeasures for preventing them. The main physiological systems will be explored before, during and after the 5 days of immersion through a battery of specific standardized tests and measurements. The objective of the study is to evaluate the physiological changes induced by 5 days of dry immersion in the female organism. The study conditions such as patient recruitment, nutrition, data collection, data management, reporting for adverse events are standardized. The results will be analyzed by scientists specializing in each field in order to better understand the dry immersion model, to compare its effects with those of the bedrest model and those of spaceflight. The clinical (adverse effects, comfort of subjects) and operational aspects are also part of the secondary objectives of the study.

Twenty healthy female subjects will participate in the study. There is no published data on dry immersion with female participation to help calculation the sample size. Moreover, female spaceflight and bedrest data are scarce, and do not provide any insight into inter-individual variability. This prolonged DI protocol in women is conceived as a pilot, descriptive, explorative study, as well as an operational and methodological study. Power-based calculation of the number of subjects is not directly applicable for such explorative studies. However, based on effect sizes obtained with previous DI studies in men, a total of 20 subjects was deemed necessary for this study.

ELIGIBILITY:
Inclusion Criteria:

* Healthy female volunteer (see below the description of medical tests and laboratory analysis performed at the selection visit),
* Age 20 to 40,
* No overweight nor excessive thinness with BMI (weight Kg/ height m2) between 20 and 26,
* Height between 158cm and 180 cm,
* Regular menstrual cycles and cycles lasting between 20 and 35 days,
* Without oestroprogestative contraception (i.e., oral progestative contraception, IUDs, implants or absence of contraception are allowed),
* Certified as healthy by a comprehensive clinical assessment (detailed medical history and complete physical examination): in particular, free from any chronic disease or any acute infectious disease or cardiovascular, neurological, ENT (especially orthostatic hypotension and vestibular disorders), orthopaedic or musculoskeletal disorders,
* Fitness level assessment:

  * if age < 35 years: 35 ml/min./kg < VO2max < 55 ml/min./kg,
  * if age > 35 years: 30 ml/min./kg < VO2max < 55 ml/min./kg,
* Non active smokers,
* No alcohol, or drug addiction, and no medical treatment (with the exception of the aforementioned accepted means of contraception),
* Covered by a Health Insurance System,
* Having signed the informed consent,
* Free from any engagement during the study.

Exclusion Criteria:

* Any history or presence of clinically relevant cardiovascular, neurological or ENT (especially orthostatic hypotension and vestibular disorders), any chronic disease; any acute infectious disease, in particular,
* Symptomatic orthostatic hypotension whatever the decrease in blood pressure,
* Asymptomatic postural hypotension defined by a decrease in SBP equal to or greater than 20 mmHg within 3 minutes when changing from the supine to the standing position,
* Cardiac rhythm disorders,
* Hypertension,
* Chronic back pains,
* Vertebral fracture, scoliosis or herniated disc,
* Glaucoma,
* Self-reported hearing problems,
* History of migraines,
* History of hiatus hernia or gastro-esophageal reflux,
* History of thyroid dysfunction, renal stones, diabetes,
* History of head trauma,
* Abnormal result for lower limbs echo-doppler,
* History of genetic muscle and bone diseases of any kind,
* Past records of thrombophlebitis, family history of thrombosis or positive response in thrombosis screening procedure (anti thrombin III, S-protein, C-protein, factor V Leiden mutation and the mutation 20210 of the prothrombin gene),
* Women who have stopped breastfeeding within 2 months before the start of the study,
* Women who have undergone an abortion within 3 months before the start of the study,
* Irregular menstrual cycles or cycles lasting less than 20 days or more than 35 days,
* Oestroprogestative contraception,
* Recent implementation or change in hormonal contraceptive (in the last 6 months),
* Bone mineral density: T-score ≤ -1.5,
* Poor tolerance to blood sampling,
* Having given whole blood (more than 8ml/kg) in a period of 8 weeks or less before the start of the experiment, or having given whole blood more than 3 times in the past year,
* Significant history of allergy, especially no dermatological allergy,
* History of food allergy,
* Significant anomaly detected in the biological analysis,
* Positive reaction to any of the following tests: HVA IgM (hepatitis A), HBs antigen (hepatitis B), anti-HVC antibodies (hepatitis C), anti-HIV1+2 antibodies,
* Vegetarian or vegan,
* Refusal to give permission to contact her general practitioner,
* Subject who, in the judgment of the investigator, is likely to be non-compliant during the study, or unable to cooperate because of a language problem or poor mental development,
* Subject already participating or in the exclusion period of a clinical research,
* Subject who has received more than 4500 Euros within 12 months for being a research subject,
* Subject who cannot be contacted in case of emergency,

MRI contraindications

* History or active claustrophobia,
* Osteosynthesis material, presence of metallic implants or any other contra-indication for MRI,
* Allergy to Gadolinium.

Vulnerable persons according to law "Code de la Santé Publique" (L1121-5 to L1121-8) :

* Pregnant women (urine pregnancy test performed at the selection visit and on the day of arrival in the facility),
* Women during childbirth and breastfeeding mothers,
* Persons deprived of their liberty by an administrative or judicial decision,
* Persons under involuntary psychiatric care,
* Persons admitted in a health or social establishment for purposes other than research,
* Minors,
* Adults subject to legal protection (subject under guardianship or trusteeship) or unable to express their consent.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2021-08-24 (Actual); Primary Completion 2021-12-08 (Actual); Study Completion 2021-12-10 (Actual)

PRIMARY OUTCOMES:
Change in orthostatic tolerance | At baseline and after five days of dry immersion
  Orthostatic tolerance will be assessed during a Lower Body Negative Pressure test (LBNP test)
Change in peak aerobic power (VO2max test) | At baseline and after five days of dry immersion
  Exercise capacity wil be assessed by graded cycling on sitting ergometer until exhaustion
Change in plasma volume | At baseline and after five days of dry immersion
  Plasma volume (L) will be assessed by the CO-rebreathing method.
Change in fluid shift distribution towards the cephalic region | At baseline, the first day to quantify the short term effect and the fifth day of dry-immersion to quantify the long term effect of fluid shift
  The hemodynamic and morphologic consequences of the fluid shift on the cephalic blood vessels (jugular vein, carotid, femoral, intracranial veins) and on the left ventricle will be investigated by ultrasound.
  The hormones involved in fluid distribution will be assessed in blood and urine samples
Change in vascular endothelium integrity | At baseline and during the five days of the dry-immersion period
  Vascular endothelium integrity will be assessed by blood parameters of vascular and endothelial integrity. Global score of endothelial state will be calculated.
Change in circadian rhythms of blood pressure | At baseline and during the five days of the dry-immersion period
  Continuous 24-h recording of blood pressure will be performed by SOMNOtouch™ NIBP system designed for ambulatory continuous measurements
Change in lower limb veins functions | At baseline, after four days of dry-immersion and after one day of recovery
  Venous compliance of lower limbs will be assessed by plethysmography.
Change in body fluid compartments by bioelectrical impedance analysis | Baseline and during five days of dry-immersion
  Extracellular, intracellular and total body water will be estimated by bioimpedance
Change in muscle strength | At baseline and after five days of dry-immersion
  Muscle strength will be assessed from single leg isometric maximal voluntary contraction on the knee extensors & flexors, the plantarflexors and dorsiflexors. The Isometric Torque will be measured in Nm. The peak of the three maximal attempts will be recorded for strength measures.
Change in muscle fatigue | At baseline and after five days of dry-immersion
  Muscle fatigability will be assessed during a submaximal isometric knee extension contraction held for 30 seconds at 50% of the baseline MVC value.
Change in muscle volume at calf level | At baseline and after five days of dry-immersion
  Muscle dehydration, eventual atrophy and fatty degeneration will be measured by quantitative Dixon MRI sequences at calf level
Change in contraction time | At baseline and after five days of dry-immersion
  Contraction time will be assessed during a tensiomyographic test in vastus lateralis, Gastrocnemius medialis and Biceps femoris of dominant leg / arm
Change in bone metabolism | At baseline, during and after 5 days of dry-immersion
  Bone metabolism in response to immobilization by dry immersion will be assessed by measuring bone biomarkers in blood samples.
Changes in cartilage metabolism | At baseline, during and after 5 days of dry-immersion
  Cartilage metabolism in response to immobilization by dry immersion will be assessed by measuring cartilage biomarkers in blood and urine samples.
Change in Resting Metabolic Rate (RMR) | At baseline, during and after 5 days of dry-immersion
  RMR will be measured by indirect calorimetry technique
Change in nitrogen balance | At baseline, during and after 5 days of dry-immersion
  Nitrogen balance is a measure of nitrogen input minus nitrogen output. Nitrogen intake is calculated with a nutrition software. Protein oxidation measured in the 24-Hour urine collection estimates nitrogen output.
Change in Body Composition measured by DEXA | At baseline and at the end of the 5 days of dry-immersion
  DEXA is a standard clinical technique to assess body composition
Change in glucose tolerance (Oral Glucose Tolerance Test) | At baseline and after 3 days of dry-immersion (to be comparable to a previous study on men)
  Glucose and insulin levels will be measured at baseline (fasting) and 30, 60, 90, and 120 minutes after drinking within 5 min a water solution containing 75 g of glucose.
Change in Core temperature | At baseline and during the 5 days of dry immersion
  Measured by electronic ingestible temperature capsules (e-Celsius Performance)
Change in height | At baseline, during and after the 5 days of dry immersion
  Measured in supine and standing position
Change in mid cerebral artery (MCA) blood flow velocity | Before and after the 5 days of dry immersion
  Transcranial Doppler measurements
Change in mood | At baseline, during and after 5 days of dry-immersion
  Change in mood is assessed using the Profile of Mood States (POMS) questionnaire. (POMS).
Change in psychological affects | At baseline, during and after 5 days of dry-immersion
  PANAS Questionnaire will be used to assess the intensity of positive and negative affective states
Change in psychological state: sleep quality | At baseline, during and after 5 days of dry-immersion
  Pittsburgh Sleep Dairy will be used to assess sleep perceived quality
Change in psychological state: mental health | At baseline, during and after 5 days of dry-immersion
  GHQ-28 Questionnaire will be used to assess psychological well-being and capture distress
Change in psychological state: coping strategies | At baseline, during and after 5 days of dry-immersion
  Brief Cope Questionnaire, designed to measure effective and ineffective ways to cope with a stressful life event, will be used to assess coping strategies
Change in cerebral autoregulation | At baseline and after 5 days of dry-immersion
  Transcranial Doppler measurements of mid cerebral artery blood flow velocity will allow to determine cerebral autoregulation
Change in Intra Cranial Pressure (ICP) | At baseline, during and after 5 days of dry-immersion
  ICP changes will be monitored through OtoAcoustic Emissions (OAE).
Change in optic nerve sheath diameter (ONSD) considered as an indirect marker for intracranial pressure (ICP) estimation. | At baseline, during and after 5 days of dry-immersion
  The optic nerve sheath diameter (ONSD) variations will be measured by echography.
Change in the optic nerve fibers thickness. | At baseline and after five days of dry-immersion
  Thickness of the optic nerve fibers will be measured by Optical Coherence Tomography (OCT)
Change in intraocular pressure (IOP) | At baseline, during and after five days of dry-immersion
  IOP measured by applanation
Change in visual acuity | At baseline and after five days of dry-immersion
  Far and near visual acuity are tested uncorrected, or if applicable with own correction with digital acuity system.
Change in visual field | At baseline and after five days of dry-immersion
  Visual field measured by standard automated perimetry
Change in the anatomical characteristics of the eye (optical biometry) | At baseline and after five days of dry-immersion
  Optical biometry measured by partial coherence interferometry
Change in the central corneal thickness | At baseline and after five days of dry-immersion
  Central corneal thickness on a single point on the cornea measured by Ultrasonic pachymetry
Change in the retina by non-mydriatic fundus retinography | At baseline and after five days of dry-immersion
  Non-mydriatic fundus retinography allows a fundus photography to be taken and thus a color image of the papilla, retinal vessels and macula.
Change in the cornea topography | At baseline and after five days of dry-immersion
  Cornea topography measured by corneal topography equipment (like Pentacam). The elevation topography according to Scheimpflug principle allows the mapping of the anterior and posterior surface of the cornea.
Change in cerebral structures and in venous circulation of the brain by MRI | At baseline and after five days of dry-immersion
  Visualization of cerebral structures and intracranial venous system will be performed by MRI coupled with injection of gadolinium.
Change in walking balance | At baseline and after five days of dry-immersion
  Walking balance will be assessed by Dynamic Gait Index, specific parameter is: total Score (range 0-24). Higher scores mean a better outcome.
Change in standing balance | At baseline and after five days of dry-immersion
  Standing balance will be assessed by posturography eyes open and eyes closed on a platform covered with 12-cm thick medium density foam.
Change in motion sickness susceptibility | At baseline and after five days of dry-immersion
  Motion Sickness Questionnaire
Change in coagulation cascade | At baseline, during and after 5 days of dry immersion
  Coagulation cascade in response to immobilization by dry immersion will be assessed by measuring coagulation parameters in blood.

CONTACTS AND LOCATIONS:
Overall Officials: Arnaud BECK, MD, Principal Investigator — MEDES - IMPS
Locations (1):
- Medes-Imps, Toulouse, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Navasiolava NM, Custaud MA, Tomilovskaya ES, Larina IM, Mano T, Gauquelin-Koch G, Gharib C, Kozlovskaya IB. Long-term dry immersion: review and prospects. Eur J Appl Physiol. 2011 Jul;111(7):1235-60. doi: 10.1007/s00421-010-1750-x. Epub 2010 Dec 14. PMID 21161267
- [Background] De Abreu S, Amirova L, Murphy R, Wallace R, Twomey L, Gauquelin-Koch G, Raverot V, Larcher F, Custaud MA, Navasiolava N. Multi-System Deconditioning in 3-Day Dry Immersion without Daily Raise. Front Physiol. 2017 Oct 13;8:799. doi: 10.3389/fphys.2017.00799. eCollection 2017. PMID 29081752
- [Background] Kermorgant M, Leca F, Nasr N, Custaud MA, Geeraerts T, Czosnyka M, Arvanitis DN, Senard JM, Pavy-Le Traon A. Impacts of Simulated Weightlessness by Dry Immersion on Optic Nerve Sheath Diameter and Cerebral Autoregulation. Front Physiol. 2017 Oct 12;8:780. doi: 10.3389/fphys.2017.00780. eCollection 2017. PMID 29075198
- [Background] Linossier MT, Amirova LE, Thomas M, Normand M, Bareille MP, Gauquelin-Koch G, Beck A, Costes-Salon MC, Bonneau C, Gharib C, Custaud MA, Vico L. Effects of short-term dry immersion on bone remodeling markers, insulin and adipokines. PLoS One. 2017 Aug 14;12(8):e0182970. doi: 10.1371/journal.pone.0182970. eCollection 2017. PMID 28806419
- [Derived] Jacob P, Robin A, Navasiolava N, Custaud MA, Ghislin S, Bareille MP, De Villemeur RB, Antunes I, Van Ombergen A, Gauquelin-Koch G, Frippiat JP. ESA VIVALDI Dry Immersion Microgravity Simulations Induce Increases in Immune Biomarkers Associated With Physical and Psychological Stress, and Sex-Specific Factors. FASEB J. 2025 Sep 15;39(17):e70993. doi: 10.1096/fj.202502198R. PMID 40892712
- [Derived] Robin A, Van Ombergen A, Laurens C, Bergouignan A, Vico L, Linossier MT, Pavy-Le Traon A, Kermorgant M, Chopard A, Py G, Green DA, Tipton M, Chouker A, Denise P, Normand H, Blanc S, Simon C, Rosnet E, Larcher F, Fernandez P, de Glisezinski I, Larrouy D, Harant-Farrugia I, Antunes I, Gauquelin-Koch G, Bareille MP, Billette De Villemeur R, Custaud MA, Navasiolava N. Comprehensive assessment of physiological responses in women during the ESA dry immersion VIVALDI microgravity simulation. Nat Commun. 2023 Oct 9;14(1):6311. doi: 10.1038/s41467-023-41990-4. PMID 37813884